CLINICAL TRIAL: NCT02854488
Title: A Global Enhanced Pharmacovigilance Pregnancy Surveillance Study of Pregnant Women Exposed to Yervoy With 5 -Year Pediatric Follow-up
Brief Title: Yervoy Pregnancy Surveillance Study
Status: Withdrawn | Type: Observational
Why Stopped: During the study period, no participants were enrolled in the study despite extensive recruitment methods.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-487
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Women Exposed to Yervoy (ipilimumab) During Pregnancy: Women Exposed to Yervoy (ipilimumab) During Pregnancy and the Children from These Pregnancies
  Interventions: Drug: Yervoy

INTERVENTIONS:
Drug: Yervoy
  Other Names: ipilimumab

SUMMARY:
The study is a global safety surveillance study of pregnancy outcomes in women who were exposed to ipilimumab during pregnancy and pediatric outcomes up to 5 years of age

ELIGIBILITY:
Inclusion Criteria:

* Documented exposure to Yervoy while pregnant or within 90 days of discontinuing treatment

Exclusion Criteria:

* Women whose ipilimumab exposure is outside the window of pregnancy exposure
* Pregnancies for which there is only paternal exposure to Yervoy

Other protocol defined inclusion/exclusion criteria could apply

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Incidence of structural birth defects in infants born to mothers exposed to Yervoy while pregnant | Birth up to 12 months
Incidence of chromosomal birth defects in infants born to mothers exposed to Yervoy while pregnant | Birth up to 12 months
Delays in developmental milestones | Birth up to 5 Years
Clinical Signs of Immune or Endocrine Dysfunction | Birth up to 5 Years
Clinical Signs of Autoimmune Disorders | Birth up to 5 Years
Clinical Signs of Serious Infections and Malignancy | Birth up to 5 Years
Adverse Pregnancy Outcomes | Time of Conception up to Birth
  Elective or spontaneous abortion, fetal death/stillbirth, pre-term delivery, ectopic or molar pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- UBC, Baltimore, Maryland, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm